CLINICAL TRIAL: NCT01933685
Title: Randomized, Double Blind Evaluation of Sequential Administration of gp120 B/E (AIDSVAX B/E) (GSID) With 1-Year Boosting in HIV-uninfected Thai Adults
Brief Title: Study of Immune Responses Induced by a HIV Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RV 328; 1939 (Other: WRAIR IRB); S-11-0005 (Other: Sponsor)
Record Dates: First submitted 2013-08-13; First posted 2013-09-02 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX B-E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIDSVAX B/E (Experimental): AIDSVAX B/E at Weeks 0, 4, 24 and 48
  Interventions: Biological: AIDSVAX B/E
- AIDSVAX B/E Placebo (Placebo Comparator): AIDSVAX B/E Placebo at Weeks 0, 4, 24 and 48
  Interventions: Biological: AIDSVAX B/E Placebo

INTERVENTIONS:
Biological: AIDSVAX B/E — 1 mL per injection (300 ug dose/antigen for a total of 600 ug/dose administered)
  Arms: AIDSVAX B/E
Biological: AIDSVAX B/E Placebo — 1 mL per injection
  Arms: AIDSVAX B/E Placebo

SUMMARY:
The purpose of this study is to define the immune responses induced by a HIV vaccine, AIDSVAX B/E. Blood and mucosal samples will be collected to assess immune responses.

DETAILED DESCRIPTION:
The primary purpose of this study is to define in HIV-uninfected volunteers the innate, cell-mediated and humoral responses induced by AIDSVAX B/E in the systemic and mucosal compartments and to characterize B cell functional specificities in peripheral blood, bone marrow and sigmoid compartments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers between age 20 and 40, available for follow up in Bangkok for a period of 18 months and having a Thai identification card.
2. Must be at low risk for HIV infection per investigator assessment.
3. Can read and write Thai language and must be able to understand and complete the informed consent process.
4. Must successfully complete a Test of Understanding (TOU) prior to enrollment.
5. Must be in good general health without clinically significant medical history.
6. HIV-uninfected per diagnostic algorithm within 45 days of enrollment.
7. Laboratory screening analysis (within normal institutional range):

   * Hemoglobin: Women >/= 12.0 g/dL, Men >/= 12.5 g/dL
   * White cell count: 4,000 to 11,000 cells/mm^3
   * Platelets: 150,000 to 450,000/mm^3
   * ALT and AST </= 1.25 institutional upper limit of reference range
   * Creatinine: </= 1.25 institutional upper limit of reference range
   * Urinalysis (dipstick) for blood and protein no greater than 1+, glucose negative
8. Female-Specific Criteria:

   * Negative human choriogonadotropin (β-HCG) urine pregnancy test for women at screening and prior to each vaccination (same day), and prior to invasive procedures.
   * Use of adequate birth control methods followed for 45 days prior to the first vaccine/placebo vaccination and will continue to be followed for at least 3 months after the final vaccine/placebo vaccination. Adequate birth control is defined as follows: Contraceptive medications delivered orally, intramuscularly, vaginally, or implanted underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), condoms, diaphragms, intrauterine device (IUD), or abstinence.

Exclusion Criteria:

1. Active, untreated syphilis
2. Asplenia: any condition resulting in the absence of a functional spleen
3. Bleeding disorder diagnosed by a medical doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), therapeutic anticoagulation resulting in an abnormal prothrombin (PT) / international normalized ration (INR) of partial prothrombin time (PTT)
4. Women breast-feeding or pregnant (positive pregnancy test) or planning to become pregnant during the window between study enrollment and 3 months after the last vaccination visit.
5. Male or female who has exchanged money or goods for sex in the last 12 months.
6. An intravenous drug user in the last 12 months.
7. History of anaphylaxis or other serious adverse reaction to vaccines any time in the past, or allergies or reactions likely to be exacerbated by any component of the vaccine or placebo, including streptomycin or neomycin.
8. Subject has received any of the following substances:

   * Chronic use of therapies that may modify immune response, such as IV immune globulin and systemic corticosteroids (in doses of >/= 20 mg/day prednisone equivalent for periods exceeding 10 days). The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least 2 weeks prior to enrollment in this study.
9. Blood products within 120 days prior to HIV screening.
10. Immunoglobulins within 30 days prior to HIV screening.
11. Any licensed vaccine within 14 days prior to initial study vaccine administration in the present study.
12. Receipt of any investigational HIV vaccine.
13. Investigational research agents or vaccine within 30 days prior to initial study vaccine administration in the present study.
14. Use of anti-tuberculosis prophylaxis or therapy during the past 90 days.
15. Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol compliance or impairs a subjects ability to give informed consent.
16. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide ideation or attempt.
17. Study site employees who are involved in the protocol and/or may have direct access to study related area.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07-03 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in Immune Response | Through Week 72
  Characterization of vaccine-induced immune responses in the systemic and mucosal compartments by intracellular cytokine staining (ICS) and IFN-gamma ELISPOT at Baseline, Weeks 4, 6, 24, 26, 48, 50 and 72.
Change in Humoral Response | Through Week 72
  Characterization of vaccine-induced humoral immune response in the systemic and mucosal compartments by binding and neutralizing antibodies at Baseline, Weeks 4, 6, 24, 26, 48, 50 and 72.

SECONDARY OUTCOMES:
Safety Monitoring | Through Week 49
  Post-vaccination reactions including erythema, induration, pain/tenderness, swelling and limitation of arm movement, fever, tiredness, chills, myalgia, arthralgia, headache, nausea, dizziness, and rash will be assessed and recorded on diary cards during the 3 days post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak,, MD, PhD, Principal Investigator — Thai Red Cross AIDS Research Centre; Jintanat Ananworanich, MD, PhD, Study Chair — US Military HIV Research Program
Locations (1):
- Thai Red Cross AIDS Research Centre, Bangkok, Thailand